CLINICAL TRIAL: NCT04310163
Title: Natural History Study Using Interview and Video Capture of Infantile and Juvenile GM1 Gangliosidosis (GM1)
Brief Title: Interviews and Video Capture in Patients With GM1 Gangliosidosis
Status: Completed | Type: Observational
Sponsor: LYSOGENE (Industry)
Collaborators: Casimir, LLC (Unknown); Cure GM1 Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: CAS-LYS003-01
Record Dates: First submitted 2020-03-12; First posted 2020-03-17 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: GM1 Gangliosidosis
Keywords: GM1 gangliosidosis; Landing disease; Lysosomal Storage Disease
MeSH Terms: conditions — Gangliosidosis, GM1; Lysosomal Storage Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Natural history — Parent interview and video capture

SUMMARY:
GM1 gangliosidosis is a rare disease for which there is a limited understanding of disease progression and meaningful outcome measures. In addition, parents report that clinic-based assessments are not always well-suited to capture all the disease features and other metrics that have an impact on the patient and family. To address the methodological challenges of this small, heterogeneous population, this study will collect patient-specific home-based video data and qualitative interviews with caregivers.

DETAILED DESCRIPTION:
This is a natural history study, for up to 2 years, during which parents or guardians of a child with GM1 gangliosidosis collect video data of patients doing specific daily life activities at baseline and follow-up timepoints throughout the study (3, 6, 12, 18, and 24 months) and/or submit videos taken in the past through a secure smart phone mobile application. The video assessments focus on several hallmarks of GM1 gangliosidosis progression. Caregivers participate in qualitative interviews to provide context for the videos and discuss any changes they observe during the study. Activity videos will be evaluated by expert clinicians using both Clinical Global Impression of Severity (CGI-S) and Clinical Global Impression of Change (CGI-C) scales. The caregiver interviews and clinician-rated activities will inform the patient-specific disease trajectories for each hallmark. There is no treatment or intervention associated with this study.

ELIGIBILITY:
Inclusion Criteria:

Be or have been the parent, legal guardian, or caretaker of a patient with GM1 gangliosidosis with:

1. Early infantile GM1 gangliosidosis
2. Late infantile GM1 gangliosidosis
3. Juvenile GM1 gangliosidosis who can walk with assistance or possesses past videos of when child could walk with assistance
4. Early or late infantile GM1 gangliosidosis who has passed away, but is in possession of videos documenting the onset and evolution of disease hallmarks of GM1 gangliosidosis

Exclusion Criteria:

GM1 gangliosidosis patient that the caregiver cares for is being treated with any experimental medication in a clinical trial setting.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population will consist of children or adolescents
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Scheduled Video Capture | up to 24 months
  Caregivers will record GM1 gangliosidosis participants doing specific activities of daily living. A list of standardized activities will be provided at baseline and the caregiver will select the activities that are relevant to the GM1 gangliosidosis participant. The activities include: gross motor skills, fine motor skills, caregiver interaction, communication, self-care and visual tracking.

SECONDARY OUTCOMES:
Unscheduled Video Capture | up to 24 months
  In addition to the scheduled video captures, spontaneously-captured videos may also be submitted by the caregivers at any time. These spontaneous videos should demonstrate any behavior or ability that the caregivers consider to be a meaningful change for the participant.
Caregiver Interviews | up to 24 months
  Casimir study staff will conduct video interviews with the caregivers at baseline and follow-up timepoints .

CONTACTS AND LOCATIONS:
Overall Officials: Mindy Leffler, MEd, Principal Investigator — Casimir Trials
Locations (1):
- Casimir Trials, Plymouth, Massachusetts, United States